CLINICAL TRIAL: NCT03822806
Title: Augmenting Patching Treatment for Amblyopia With Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erick D. Bothun, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-010474
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Exercise in addition to Patching (Experimental): Patch for 2 hours a day, and exercise (using the videogame JustDance) for the first 30 minutes of those 2 hours using the video game (continuing to wear the patch for 90 minutes after exercise).
  Interventions: Other: Physical Exercise in addition to Patching

INTERVENTIONS:
Other: Physical Exercise in addition to Patching — Patch for 2 hours a day, and exercise for the first 30 minutes of those 2 hours using the video game

SUMMARY:
Researches are trying to establish whether moderate exercise enhances the treatment benefit of patching 2 hours a day for residual amblyopia in children.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 to < 17 years old
* Cycloplegic refraction within past year
* Diagnosis of residual amblyopia, with no evidence of regression of amblyopic eye visual acuity by 1 or more LogMAR from best previous
* Completed at least 6 months prior patching treatment (minimum 2 hours/day) or atropine treatment.
* Stable visual acuity as defined by <1 LogMAR change over 2 visits
* Xbox 360 Kinect, Wii or WiiU gaming system in the home, or a different gaming system with a version of Just Dance® already in the home.

Exclusion Criteria:

* Known problems with exercise tolerance
* No gaming system in the home that supports Just Dance® Kids 2014, and no existing version of Just Dance® in the home
* Current atropine treatment for amblyopia

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1 month (3 weeks to 8 weeks) after initiating game play
  The primary outcome measure will be LogMAR visual acuity measured 1 month (primary analysis window 3 weeks to 8 weeks) after initiating game play.

CONTACTS AND LOCATIONS:
Overall Officials: Erick Bothun, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials